CLINICAL TRIAL: NCT03417310
Title: Studying the Clinical Applications of "H" Joystick for Reduction in Femoral Shaft Fractures
Brief Title: Clinical Applications of a Joystick in Femoral Shaft Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, John Wong, Assistant Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015030024
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Femur Shaft Fracture
Keywords: closed reduction; locked intramedullary nailing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "H" joystick (Experimental): Patients are treated with the "H" joystick on a traction table
  Interventions: Device: "H" joystick
- Common reduction methods (Active Comparator): Patients are treated with common reduction methods on a traction table
  Interventions: Procedure: Common reduction methods

INTERVENTIONS:
Device: "H" joystick — A joystick that corrects lateral displacement and angulation for multi-direction reduction
  Arms: "H" joystick
Procedure: Common reduction methods — Manual reduction methods without the assistance of any devices
  Arms: Common reduction methods

SUMMARY:
This study will use a new "H" joystick for reduction on patients with femur fractures to investigate the reduction time, operating time and bone healing status for the evaluation of the clinical application benefits of this joystick.

DETAILED DESCRIPTION:
This study will design a new "H" joystick for reduction (which has received the national utility model patent) and will use this equipment on 80 patients (55 males, 25 females) with femur fractures to investigate the reduction time, operating time and bone healing status for the evaluation of the clinical application benefits of this joystick.

ELIGIBILITY:
Inclusion Criteria:

* Femur shaft fractures

Exclusion Criteria:

* Not suitable to receive intramedullary nail treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Operating time | One day
  Duration of operation
Fluoroscopy times | One day
  The number of times for fluoroscopy
Blood loss | One day
  The amount of blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Xinjia Hu, MD, PhD, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No